CLINICAL TRIAL: NCT04927208
Title: Effect of Essential Aminoacid Supplementation and Exercise on Skeletal Muscle Function in Hemodialysis Patients
Brief Title: Effect of Exercise and Protein Supplementation on Muscle Function in Patients With Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-ED-2021-001
Record Dates: First submitted 2021-05-17; First posted 2021-06-15 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise; Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improved skeletal muscle function due to protein supplementation (Experimental): Experimental: Intervention group Improved skeletal muscle function due to protein supplementation
  Interventions: Other: exercise and nutritional support

INTERVENTIONS:
Other: exercise and nutritional support — resistance exercise and protein supplementation including branched chain amino acids for 12 weeks
  Other: Combined exercise and nutrition intervention resistance exercise and nutritional supplementation for 12 weeks

SUMMARY:
Sarcopenia can be easily observed in patients with hemodialysis. However, there were few studies on the precise concept and diagnostic criteria for sarcopenia in patients with hemodialysis. The investigators have already recognized the sarcopenia-associated mortality and morbidity in patients with hemodialysis. However, intervention studies on hemodialysis patients with sarcopenia have not been conducted until now. Here, The investigators aim a pilot study to evaluate the effectiveness of the combined exercise and nutrition intervention for sarcopenia in patients with hemodialysis.

This is a prospective study with 60 patients with hemodialysis who were diagnosed as sarcopenia or frailty in our previous cohort study. Combined intervention will consist of resistance exercise and nutritional supplementation for 12 weeks. The primary outcome of this study is muscle mass and handgrip strength after 12 weeks' intervention. All functional outcomes will be measured at 0, 12, and 24 weeks after intervention. The data will be analysed using the intention-to-treat principle.

DETAILED DESCRIPTION:
While feasible, inexpensive, and non radiation-exposed tools such as bioimpedance analysis have been used to measure appendicular skeletal muscle mass. In addition, isokinetic strength will be measured by a dynamometer for hand grip strength to evaluate sarcopenia. The main two axes of treatment of conventional sarcopenia are muscle resistance exercises and protein supplementation including branched chain amino acids. Therefore, it is necessary to confirm the clinical effect by intervention for resistance exercise and nutritional supplementation in patients with hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemodialysis
* Community-dwellers
* Able to walk with or without assistive devices for more than 100 meters

Exclusion Criteria:

* A person with cancer disease.
* People with psychiatric symptoms.
* A person who has an absorption disorder or has a history of resection of the small intestine or colon
* Pregnant women
* A person treated for acute bacterial infections
* A person who is in a wheelchair due to inconvenience in walking.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Handgrip strength in Kg | 24weeks
  Measurement of handle strength using a portable dynamometer to view the function of skeletal muscle.

SECONDARY OUTCOMES:
The total score of SPPB(Short Physical Performance Battery) | 24 weeks
  The total score is the sum of 5 times CST score and balance test score and gait speed test score for 4meter.
The second of 5 times Chair Stand Test | 24 weeks
  Pre test, participants fold their arms across their chest and try to stand up once from a chair. And Measures the time required to perform five rises from a chair to an upright position as fast as possible without the use of the arms.
skeletal muscle mass index in cm2/m2 | 24 weeks
  The SMI was calculated according to the following formula: skeletal muscle mass (cm 2) / height 2 (m 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Ju SH, Lee EJ, Sim BC, Nga HT, Lee HY, Tian J, Cho KJ, Park H, Choi DE, Ham YR, Yi HS. Leucine-enriched amino acid supplementation and exercise to prevent sarcopenia in patients on hemodialysis: a single-arm pilot study. Front Nutr. 2023 Apr 28;10:1069651. doi: 10.3389/fnut.2023.1069651. eCollection 2023. PMID 37187878